CLINICAL TRIAL: NCT00212472
Title: An International Randomised Controlled Trial Of Immune Tolerance Induction
Brief Title: International Immune Tolerance Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The DSMB recommended stopping the study due to safety concerns.
Sponsor: New York Presbyterian Hospital (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Donna DiMichele, MD, New York Presbyterian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITI
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-10

CONDITIONS: Hemophilia A With Inhibitors
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Low-dose treatment (50 FVIII u/kg three times a week).
  Interventions: Drug: Factor VIII concentrates; Other: Low-dose treatment
- 2 (Active Comparator): High-dose treatment (200 FVIII u/kg per day).
  Interventions: Drug: Factor VIII concentrates; Other: High-dose treatment

INTERVENTIONS:
Drug: Factor VIII concentrates — To be determined at the discretion of the investigator.
Other: Low-dose treatment — 50 FVIII u/kg three times a week.
  Arms: 1
Other: High-dose treatment — 200 FVIII u/kg per day.
  Arms: 2

SUMMARY:
The purpose of this study is to see if a low-dose arm or a high dose-arm of immune tolerance is more effective in eliminating inhibitors in patients with hemophilia A.

DETAILED DESCRIPTION:
Subjects will be randomized into a low-dose or high-dose immune tolerance regimen and this study will compare the success rates, the time to achieve tolerance,the complications and the cost of both regimens.It will also aim to identify predictors of successful immune tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (FVIII level <1%).
* A maximum historical inhibitor titer of between 5 BU and 200 BU that must be confirmed once prior to the beginning of ITI.
* The inhibitor titer should be <10 BU at the start of ITI, confirmed once.
* The inhibitor must be present for <24 months when ITI begins.
* Maximum age of 7 at the start of ITI.
* Willingness to comply with the protocol.

Exclusion Criteria:

* Moderate or mild hemophilia A (FVIII level >1%).
* Spontaneous disappearance of the inhibitor prior to ITI.
* Historical maximum inhibitor titer <5 BU or > 200 BU before starting ITI.
* Inhibitor titer > 10 BU at the start of ITI.
* Inhibitor present for more than 24 months before starting ITI.
* Systemic immunomodulatory drug therapy during immune tolerance e.g. corticosteroids (< 5 days every 2 months maximum dose 2 mg/kg or 60 mg/day), azathioprine, cyclophosphamide, high-dose immunoglobulin or the use of a protein A column or plasmapheresis.
* Age > 7 years at the start of ITI.
* Inability or unwillingness to comply with the protocol.
* Previous attempt at ITI.

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2002-07; Primary Completion 2010-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Success-rate and partial success-rate | Up to 69 months
The time from the start of ITI to successful tolerance | Up to 33 months
The comparative cost-effectiveness of the two treatment arms | Up to 69 months
A comparative assessment of morbidity between the two treatment arms including: number of intercurrent bleeds, infections and number of hospital in-patient days. | Up to 69 months
The inhibitor recurrence (relapse) rate in the first twelve months after successful ITI. | Up to 45 months

SECONDARY OUTCOMES:
The dose-regimen, success rate and time to ITI, | Up to 69 months
The starting inhibitor titre, success rate and time to ITI, | Up to 69 months
The peak historical inhibitor titre, success rate and time to ITI, | Up to 69 months
The peak inhibitor titre after starting ITI, success rate and time to success, | Up to 69 months
The age at the time of inhibitor detection, success-rate and time to success, | Up to 69 months
The number of factor VIII treatment days between inhibitor detection and initiation of ITI, success of ITI. | Up to 69 months
The type of concentrate used (von Willebrand factor-containing, monoclonal or recombinant), success rate and time to success, | Up to 69 months
The effect of interim infections/immunisations, success rate and time to success, | Up to 69 months
The effect of treatment interruption, success rate and time to success. | Up to 69 months

CONTACTS AND LOCATIONS:
Overall Officials: Donna M DiMichele, MD, Principal Investigator — Weill Cornell Medical College-NY Presybetrian Hospital; Charles Hay, MD, Principal Investigator — Manchester Royal Infirmary
Locations (39):
- United States (39):
  - University of Alabama Birmingham Medical Center, Birmingham, Alabama
  - City of Hope Medical Center, Duarte, California
  - Children's Hospital of Orange County, Orange, California
  - Mountain States Regional Hemophilia and Thrombosis Center, Aurora, Colorado
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Rush Presbyterian St. Lukes, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Comprehensive Bleeding Disorders Center, Peoria, Illinois
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan Health Hospitals, Ann Arbor, Michigan
  - MSU Centers for Bleeding & Clotting Disorders, East Lansing, Michigan
  - Children's Hospital Minneapolis, Minneapolis, Minnesota
  - Mayo Comprehensive Hemophilia Center, Rochester, Minnesota
  - Kansas City Regional Hemophilia Center-The Children's Mercy Hospital, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Ted R. Montoya Hemophilia Treatment Center, Albuquerque, New Mexico
  - NY Presbyterian Hospital, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Section of Hem/Onc, Philadelphia, Pennsylvania
  - The Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center-Gulf States Hemophilia & Thrombosis Center, Houston, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Virginia
  - Comprehensive Center for Bleeding Disorders, Milwaukee, Wisconsin